CLINICAL TRIAL: NCT04963452
Title: Does Body Mass Index Impact the Outcome of Dural Puncture Epidural in Parturients Undergoing Normal Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: R 149/2021
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; Labor Pain
MeSH Terms: conditions — Obesity, Morbid; Labor Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): Normal weight BMI 20-24.9 kg/m2
  Interventions: Other: Dural puncture epidural
- Group 2 (Active Comparator): Morbid Obese BMI : 40-49.9 kg/m2
  Interventions: Other: Dural puncture epidural

INTERVENTIONS:
Other: Dural puncture epidural — Parturients, between 18 and 45 years of age, with cervical dilation less than 5 cm were consented to receive a DPE technique, with a single dural puncture with a 26-gauge spinal needle. After successful placement of the epidural catheter and puncturing the dura; 20 mL of bupivacaine 0.25% was administered through the epidural catheter and a patient-controlled epidural infusion of bupivacaine was initiated.

SUMMARY:
Recently, the dural puncture epidural (DPE) technique has emerged as a novel method of labor analgesia. The DPE technique is a modification of the combined spinal epidural (CSE) technique, where a dural perforation is created from a spinal needle but intrathecal medication administration is withheld. The DPE technique has been shown to improve caudal spread of analgesia compared with epidural technique without the side effects observed with the CSE technique.

DETAILED DESCRIPTION:
Investigators designed this prospective interventional study to determine if morbid obesity would influence DPE technique regarding labor analgesia onset and block characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 45 years old,
2. Physical status American society of anesthesiology (ASA) II,
3. Singleton,
4. Vertex fetuses at 37-41 weeks' gestation,
5. Nulliparous and multiparous women,
6. Immediately before epidural placement, subjects marked a VNRS score during an active contraction and parturients with VNRS ≥ 50 were included
7. Cervical dilatation < 5 cm

Exclusion Criteria:

1. Contraindications to regional anesthesia
2. Refuse to participate
3. No pain
4. Severe systemic disease (kidney, liver, pulmonary, endocrine, cardiac)
5. Conditions associated with an increased risk of a cesarean delivery (i.e., history of uterine anomaly or surgery) and vaginal birth after cesarean delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturients undergoing normal vaginal delivery
Enrollment: 64 (Actual)
Dates: Start 2021-08-29 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adequate analgesia | 5 minutes
  The primary outcome of this study is the incidence of patients having adequate analgesia (VNRS <30) at 5 minutes of epidural activation

SECONDARY OUTCOMES:
Verbal numerical pain score scale ( 0 being no pain and 100 being the worst pain ) | 6 hours
  Verbal numerical pain score (VNRS) (pain) was recorded before epidural (0 min baseline), at 5 min, 10 min, 15 min and then every 15 min till 1 hour and then every 30 min till delivery.
Sensory level of DPE by pricking by blunt head of a pin | 6 hours
  * Was recorded before epidural (0 min-baseline), at 5 min, 10 min, 15 min and then every 15 min till 1 hour and then every 30 min till delivery.
  * Sensory level of DPE was assessed by loss of sensation to prick by blunt head of a pin.
Motor block Bromage score (1 being complete motor block and 6 being no motor block) | 6 hours
  * Motor strength was assessed with a modified Bromage score
  * Was recorded before epidural (0 min baseline), at 5 min, 10 min, 15 min and then every 15 min till 1 hour and then every 30 min till delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No